CLINICAL TRIAL: NCT06430931
Title: Biological OviTex Versus Synthetic Graft in Robotic Prolapse Surgery: a Multicentre, Phase 11-111, Partially Randomised Patient Preference Trial
Brief Title: Biological OviTex Versus Synthetic Graft in Robotic Prolapse Surgery
Acronym: ProTex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meander Medical Center (Other)
Collaborators: Health Holland (Other)
Responsible Party: Principal Investigator, Esther Consten, Clinical Professor, Meander Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79184.100.22
Record Dates: First submitted 2024-05-02; First posted 2024-05-28 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Disorders; Prolapse; Prolapse Rectal; Prolapse Genital; Prolapse Pelvic; Rectocele; Prolapse Uterus; Cystocele; Enterocele; Prolapse Bladder; Prolapse; Cervix
Keywords: Prolapse; Abdominal prolapse Surgery; Biological mesh; OviTex; VMR; sacrocolporectopexy
MeSH Terms: conditions — Prolapse; Rectal Prolapse; Rectocele; Uterine Prolapse; Cystocele; Hernia

STUDY DESIGN:
Intervention Model Description: Multi-centre prospective non-inferior patient-preference study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Polypropylene mesh (Active Comparator): Polypropylene mesh (Prolene, PMN3, Ethicon Inc Johnson & Johnson, Amersfoort, The Netherlands; weight 78 g/m2)
  Interventions: Procedure: Minimal invasive abdominal prolapse surgery using Polypropylene mesh
- OviTex 1S permanent mesh (Experimental): OviTex Reinforced BioScaffold, Permanent Polymer composed of ovine (sheep) forestomach extracellular matrix (ECM) and polypropylene.
  Interventions: Procedure: Minimal invasive abdominal prolapse surgery using OviTex 1S permanent mesh

INTERVENTIONS:
Procedure: Minimal invasive abdominal prolapse surgery using Polypropylene mesh — All procedures will be performed with robotic assistance of the da Vinci Si-HD (intuitive Surgical, Inc, Sunnyvale, CA).
  Other Names: Ventral mesh rectopexy; Sacrocolporectopexy
  Arms: Polypropylene mesh
Procedure: Minimal invasive abdominal prolapse surgery using OviTex 1S permanent mesh — All procedures will be performed with robotic assistance of the da Vinci Si-HD (intuitive Surgical, Inc, Sunnyvale, CA).
  Other Names: Ventral mesh rectopexy; Sacrocolporectopexy
  Arms: OviTex 1S permanent mesh

SUMMARY:
This prospective study aims to assess the efficacy of the OviTex 1S permanent mesh in pelvic floor surgery in comparison with the current standard polypropylene mesh.

DETAILED DESCRIPTION:
Minimal-invasive ventral mesh rectopexy (VMR) and sacrocolporectopexy (SCR) or cervicopexy are widely accepted treatments for patients suffering from pelvic prolapse. Choice of material used in VMR or SCRP - synthetic or biologic surgical mesh - remains subject of debate. Recent ban in the usage of non abdominal but transvaginal, mesh for pelvic organ prolapse (POP) in April 2019, by the Food and Drug Administration (FDA) has negatively influenced the perception on all sorts of surgical mesh. Currently, the most widely used mesh in VMR is synthetic and has shown good results regarding recurrence, mesh exposure and functional outcome. Although complication rates are low, the serious complications of fistulation, exposition, and dyspareunia are reasons to opt for a more expensive biological mesh. High-quality evidence of synthetic versus biological mesh is lacking, which does not stop resistance against synthetic mesh from growing. This has even led to concerns and questions about synthetic mesh use from the Dutch government addressed at the medical professionals and options for alternatives are being asked.

Biological grafts are characterized by degradation of the implant and regeneration of host tissue. It is assumed that this process of degradation and remodeling decreases the risk of exposition and infection. However, this transformation may possibly lead to a higher chance of recurrence in the long term. Rate of recurrence, but also graft-related complications (GRC) to a lesser extent, largely depends on duration of follow-up. Since biological graft implementation in VMR and SCR is relatively new and its usage is restricted due to higher costs, evidence on biological mesh with long term follow-up is limited. In addition, there is a significant difference in various described biological meshes. This is important to keep in mind when comparing outcome of VMR or SCR with synthetic versus biologic mesh.

In VMR there are no randomised controlled trials on synthetic versus biological mesh. The biological meshes studied thus far are Biodesign and Permacol. Mesh exposure rates after VMR with Biodesign and Permacol have both been studied in three studies in total (N = 349 and N = 425 in total respectively) and show low mesh exposure rates of 0 to 0.1%. In comparison, GRC after VMR with synthetic non-resorbable mesh (like polypropylene) are around 2%. Recurrence rates after synthetic mesh in VMR range between 2% and 14% after a median follow-up of 12-61 months. When comparing studies on biologic implants that report on recurrence rates there seems to be a slight difference in favor of Biodesign. Studies on Biodesign in VMR with a median follow-up ranging between 12 and 47 months show a recurrence rate around 5%. Literature on Permacol shows higher recurrence rates ranging between 5 to 14% after a median follow-up of 12 to 29 months.

In sacrocolpopexy (SCP) allografts and xenografts have been investigated as an alternative for polypropylene. A randomised controlled trial compared SCP using polypropylene mesh with solvent cadaveric fascia lata. After one year of follow-up, polypropylene mesh had a higher anatomical cure rate than cadaveric fascia lata (91 percent versus 68 percent; p=0.007). Two GRC occurred in patients who received polypropylene mesh, while none occurred in the allograft group (p= 0.5). Another RCT with the same comparison and a follow-up of 5 years showed similar results, with considering cadaveric fascia not as strong of a support. Deprest et al. compared polypropylene mesh with porcine grafts in a prospective study and found xenografts to be associated with more apical failures and reoperations than with a polypropylene mesh (21 percent versus 3 percent; p = 0.01).However, there was no significant difference in functional outcomes between the two groups. An exposure rate of 11 percent was described in both groups. A more recent study concluded, by analyzing clinical outcomes and patients satisfaction, that a non-crosslinked ADM patch can be a good alternative to synthetic polypropylene mesh in patients undergoing SCP.

Although Biodesign (Surgisis), Permacol and other are all grouped under the common denominator 'Biologic mesh', each of these products is unique. There are differences in tissue source, differences in the processes used to decellularize the tissue and differences in the final processing steps such as sterilization and preservation. As a result, there are significant variations in biological and clinical performance between these products. Permacol, which is purposely cross-linked pig dermis, behaves like a synthetic material in-vivo and induces a permanent foreign body response, leading to encapsulation. This prevents integration with and in the surrounding tissue. Consequently, high rates of mesh exposure occur with Permacol implants. Biodesign, one of the early biologics, is derived from small intestinal submucosa and is a non-cross-linked mesh. Likely due to its (proprietary) processing, Biodesign in practice often dissolves before healing and remodeling can take place.

A novelty on the surgical mesh market is OviTex. It is produced by Aroa Biosurgery and consist of sterile sheep extracellular matrix (ECM) interwoven with a (absorbable or non-absorbable) synthetic fiber. OviTex comes with a grid of absorbable polyglycolic acid (PGA) or permanent polypropylene and with differing amounts of layers (Core, 1S and 2S). Unique to OviTex is its composition, which consists of essential components required for regeneration of host tissue. Additionally, the coupling of an ECM with a (absorbable) synthetic fiber provide strength without the need to cross-link the ECM. Moreover, OviTex is lower in costs than any other biological mesh on the market. Since the use of synthetic meshes in pelvic floor surgery has come under scrutiny, patients are tempted to undergo a resection rectopexy as an alternative to VMR with polypropylene. Apart from the fact that the resection is associated with a higher risk of complications due to the application of an anastomosis, the recovery time is much longer. The hospitalization period would be longer and therefore the costs compared to prolapse surgery with OviTex would be higher.

Preliminary results of a recent pilot study at Meander MC showed that the use of an OviTex PGA (with absorbable grid) mesh in the pelvic floor is feasible and safe. Nevertheless, 2 out of 11 patients who completed follow-up of 6 months showed an early anatomical recurrence. This suggests that the use of permanent synthetic fiber may be necessary for a more durable repair and fewer recurrences than using OviTex PGA. Although resistance against synthetic grafts is growing, OviTex Permanent contains 96% sheep ECM and only 4% polymer, compared to the standard Prolene mesh which is 100% polymer (polymer areal density 16g/m2 OviTex 1S vs. 76g/m2 prolene). Furthermore, the polymer is embedded in the ECM which further attenuates any inflammatory response. Observations in primates show that the minimized amount of embedded synthetic reinforcement results in an implant that, histologically, behaves like a biologic mesh yet maintains its functional structure. This is the first prospective multicenter study using a OviTex 1S mesh. Although the material ovine was studies before, little is known about the feasibility of enrolling these patients into randomised studies in the Netherlands and about the feasibility, safety, and tolerance of the OviTex 1s is this setting. Therefore, the investigators decided to start with a phase II study. This allows for adequate monitoring of the feasibility, safety, and tolerance of the experimental treatment.

There are no studies comparing OviTex to the current standard (Prolene, PMN3, Ethicon Inc Johnson & Johnson, Amersfoort, The Netherlands) Therefore, a comparative study should be conducted before OviTex is used as a biologic alternative for polypropylene in VMR on a larger scale. Following the OviTex pilot study, the investigators aim to conduct a follow-up study (ProTex trial) in which, both in the short and longer term, the efficacy of the OviTex mesh in pelvic floor surgery will be assessed in comparison with the current standard polypropylene, by means of a non-inferiority test.

ELIGIBILITY:
Inclusion Criteria:

* Indication for VMR or SCR set by the treating surgeon/gynecologist in accordance to the current guidelines on rectal and pelvic prolapse;
* Counselled for therapeutic options and given informed consent for VMR or SCR;
* Counselled for different types of mesh (OviTex or Prolene) and randomisation;
* Written informed consent for randomisation, OviTex implant or Prolene;
* Written informed consent for observational data collection.

Exclusion Criteria:

* Mentally incompetent patients (unable to fulfil questionnaires).
* Allergy to ovine rumen.
* A medical history of pelvic radiation therapy.
* Scheduled for a redo-rectopexy.
* A medical history of previously implanted pelvic floor meshes or native tissue.
* Language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Main study parameter/endpoint phase II: rate of complications | 90days postoperative
  Post-operative complications. The Clavien Dindo Classification is used to rank the severity of a surgical complication
Main study parameter/endpoint phase ll: number of participants with post-operative morbidity | 90days postoperative
  Post-operative morbidity measured by reoperations, reinterventions, readmissions,
Main study parameter/endpoint phase Ill: Pelvic Floor Distress lnventory-20 score (PFDl-20) | 24 months postoperative
  Constipation, incontinence and urogenital functioning (questionnaire, validated scoring system: Pelvic Floor Distress lnventory-20 (PFDl-20). The Pelvic Floor Distress Inventory-20 (PFDI-20) is a questionnaire used to assess the presence and severity of symptoms related to pelvic floor disorders. The PFDI-20 consists of 20 questions divided into three subscales: the Pelvic Organ Prolapse Distress Inventory (POPDI), the Colorectal-Anal Distress Inventory (CRADI), and the Urinary Distress Inventory (UDI).
  Scale Details:
  Minimum Score: 0 Maximum Score: 300 Interpretation: Higher scores indicate a worse outcome, reflecting greater distress or more severe symptoms.

SECONDARY OUTCOMES:
Constipation | 24 months postoperative
  Questionnaire, validated scoring system: Altomare obstructive defecation score (ODS) with a maximum score of 31. A higher score on the Altomare scale indicates a greater severity of constipation. Scores will be compared before and after treatment.
Incontinence | 24 months postoperative
  Questionnaire, validated scoring system: Fecal Incontinence Severity Index (FISI) with a maximum score of 60. A higher FISI score indicates more severe fecal incontinence. Scores will be compared before and after treatment.
Quality of life (Qol) pre- and postoperatively by the Patient Global Impression of Improvement (PGl-I). | 24 months postoperative
  Objectified primarily by the Patient Global Impression of Improvement (PGl-I). The PGI-I scale measures the patient's perception of improvement (or lack thereof) in their condition following treatment. 1 - Very much improved: Significant improvement in condition.
  2 - Much improved: Noticeable improvement in condition. 3 - Minimally improved: Slight improvement in condition. 4 - No change: Condition has not changed. 5 - Minimally worse: Slight worsening of condition. 6 - Much worse: Noticeable worsening of condition. 7 - Very much worse: Significant worsening of condition.
Quality of life (Qol) pre- and postoperatively by the Patient Global Impression of Severity (PGl-S). | 24 months postoperative
  Objectified primarily by the Patient Global Impression of Severity (PGl-S). The PGI-S scale measures the patient's perception of the severity of their condition at a specific point in time. 1 - Normal: No symptoms.
  2 - Borderline: Barely noticeable symptoms. 3 - Mild: Symptoms are present but do not significantly interfere with daily activities.
  4 - Moderate: Symptoms are more noticeable and do interfere with daily activities.
  5 - Severe: Symptoms are significant and very disruptive to daily activities. 6 - Very severe: Symptoms are extremely disruptive and may prevent daily activities.
  7 - Extremely severe: Symptoms are debilitating.
Quality of life (Qol) pre- and postoperatively by the European Quality of Life Five Dimension (EQ-5D). | 24 months postoperative
  Objectified primarily by the European Quality of Life Five Dimension (EQ-5D). The European Quality of Life Five Dimension (EQ-5D) measures health-related quality of life using a descriptive system with five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) rated at three severity levels, and an EQ visual analogue scale (EQ VAS) from 0 to 100 for overall health perception.
Quality of life (Qol) pre- and postoperatively by the Pelvic Floor impact Questionnaire (PFIQ-7) | 24 months postoperative
  Objectified primarily by the Pelvic Floor impact Questionnaire (PFIQ-7). Higher scores on the PFIQ-7 indicate a greater negative impact of pelvic floor disorders on the patient's quality of life.
Number of patients with post-operative morbidity | 24 months postoperative
  Measured by reoperations, reinterventions, readmissions, and serious adverse advents.
Number of patients with anatomic recurrence of the rectal prolapse | 24 months postoperative
  Measured by defecogram or MR defecography in rest and during Valsalva maneuver.
Rate of rectal prolapse recurrence and complications | 24 months postoperative
  Complaints, physical examination, addition research, re-operation and readmission
Number of patients with anatomic recurrence of pelvic organ prolapse (POP) | 24 months postoperative
  Using the simplified Pelvic Organ Prolapse Quantification (sPOPQ)
Sexual functioning pre- and postoperatively scores on the PSIQ-IR | 24 months postoperative
  By the questionnaire Prolapse Incontinence Sexual Inventory Questionnaire (PSIQ-IR). Lower Scores: Indicate greater sexual dysfunction and more issues related to the conditions.
Length of hospital stay in days | 24 months postoperative
Rate of extra outpatient visits because of complaints | 24 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Esther Consten, Prof.dr, Principal Investigator — Meander Medisch Centrum
Locations (1):
- Meander Medisch Centrum, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request after publication of the primary study results. Data will be available for academic research purposes, subject to approval of a research proposal and a data sharing agreement. Requests should be addressed to the principal investigator.
Supporting Information: Study Protocol
Time Frame: After publication of the primary study results.